CLINICAL TRIAL: NCT06622720
Title: Laparoscopic Elective Colorectal Procedures Performed by Supervised Residents Are Safe and Sufficient.
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Zofia Orzeszko, MD, Jagiellonian University
Other Study IDs: 2024.000.463
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Surgical Training; Residency
Keywords: Colorectal Cancer; Surgical Training; Residency; Colorectal Surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Residents: Individuals undergoing elective colorectal resection due to cancer performed by residents between January 2022 and December 2023.
  Interventions: Procedure: surgery
- Colorectal surgeons: Individuals undergoing elective colorectal resection due to cancer performed by experienced colorectal surgeons between January 2022 and December 2023.
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — The colorectal surgery of any type conducted in any approach in the timeframe

SUMMARY:
The ability to perform laparoscopic colorectal surgery is an essential attribute of a general surgeon. Data on the participation of residents and the outcomes of colorectal procedures performed by surgeons in training are in demand. The objective of this study is to comprehensively investigate the outcomes of colorectal procedures performed by general surgery residents supervised by experienced colorectal surgeons and assess their previous laparoscopic experience.

DETAILED DESCRIPTION:
The ability to perform laparoscopic colorectal surgery is an essential attribute of a general surgeon. Residents' contribution to colorectal procedures ranges from 33 to 40%. Few papers describe the outcomes of treatment provided by residents. The learning curve in colorectal techniques requires 88 to 152 cases to reach proficiency. Data on the participation of residents and the outcomes of procedures performed by surgeons in training are in demand. The objective of this study is to comprehensively investigate the outcomes of colorectal procedures performed by general surgery residents supervised by experienced colorectal surgeons and assess their previous laparoscopic experience. A retrospective single-center analysis was performed based on a review of database records. It included 498 elective colorectal procedures performed in a high-volume colorectal surgery center, where over 200 procedures are performed each year. The study included all individuals undergoing elective colorectal resection due to cancer between January 2022 and December 2023. 43 procedures were performed by residents and 455 by experienced colorectal surgeons. The procedures were performed by five experienced colorectal surgeons and three residents in their third to sixth year of surgical training. When performing evaluated procedures, residents were performed under the surveillance of experienced colorectal surgeons, according to Polish law requirements.

ELIGIBILITY:
Inclusion Criteria:

* all individuals undergoing elective colorectal resection due to cancer between January 2022 and December 2023 in a single colorectal center.

Exclusion Criteria:

* stoma creation
* a history of inflammatory bowel disease
* a history of bowel resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included all adult individuals undergoing elective colorectal resection due to cancer between January 2022 and December 2023 in a single colorectal center.
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of complete resections | 1st January 2021 - 31th December 2023
  Resection is noted as complete (R0) when resection margins are clear from cancer infiltration microscopically and macroscopically.
The number of resected lymph nodes | 1st January 2021 - 31th December 2023
  Reported number of lymph nodes in histopathological result
The duration of surgery | 1st January 2021 - 31th December 2023
  Reported surgery time
The length of hospital stay | 1st January 2021 - 31th December 2023
  Reported days in hospital

SECONDARY OUTCOMES:
The rate of readmissions | 1st January 2021 - 31th December 2023
  Reported number of readmissions
The rate of anastomosis leaks | 1st January 2021 - 31th December 2023
  Reported number of anastomosis leaks
The rate of postoperative ileus | 1st January 2021 - 31th December 2023
  Reported number of postoperative ileus
The rate of reoperations | 1st January 2021 - 31th December 2023
  The number of reoperations at any cause associated with primary surgery (both surgical and endoscopic interventions).
The rate of surgical site infection | 1st January 2021 - 31th December 2023
  Reported number of surgical site infection
Mortality | 1st January 2021 - 31th December 2023
  Reported mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mirosław Szura, Prof, PhD, Study Chair — Jagiellonian University
Locations (1):
- Hospital of St John of God, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
The data will not be shared.

REFERENCES:
- [Background] Ofshteyn A, Terry M, Bingmer K, Stein SL, Steinhagen E. General surgery resident experience with anorectal surgery. Am J Surg. 2020 Jun;219(6):993-997. doi: 10.1016/j.amjsurg.2019.08.010. Epub 2019 Aug 17. PMID 31445669
- [Background] Saraidaridis JT, Read TE, Marcello PW, Schoetz DJ, Rusin LC, Kleiman DA, Melnitchouk N, Roberts PL, Breen EM. What do Young Colorectal Surgeons Value From Their CRS Residency Training? J Surg Educ. 2019 May-Jun;76(3):720-726. doi: 10.1016/j.jsurg.2018.09.013. Epub 2018 Oct 17. PMID 30342854
- [Background] Bustamante Recuenco C, Alonso-Lamberti Rizo L, Salazar Carrasco A, Valle Rubio A, Cendrero Martin M, Jimenez Carneros V, Ramos Rodriguez JL, Jimenez Miramon FJ. Resident training in colorectal laparoscopic surgery: A retrospective morbidity, mortality and survival analysis of 408 cases in our environment. Cir Esp (Engl Ed). 2022 Sep;100(9):555-561. doi: 10.1016/j.cireng.2022.06.016. Epub 2022 Jun 11. PMID 35697242
- [Background] Nijhof HW, Silvis R, Vuylsteke RCLM, Oosterling SJ, Rijna H, Stockmann HBAC. Training residents in laparoscopic colorectal surgery: is supervised surgery safe? Surg Endosc. 2017 Jun;31(6):2602-2606. doi: 10.1007/s00464-016-5268-0. Epub 2016 Oct 4. PMID 27704242
- [Background] Miskovic D, Ni M, Wyles SM, Tekkis P, Hanna GB. Learning curve and case selection in laparoscopic colorectal surgery: systematic review and international multicenter analysis of 4852 cases. Dis Colon Rectum. 2012 Dec;55(12):1300-10. doi: 10.1097/DCR.0b013e31826ab4dd. PMID 23135590
- [Background] Perivoliotis K, Baloyiannis I, Mamaloudis I, Volakakis G, Valaroutsos A, Tzovaras G. Change point analysis validation of the learning curve in laparoscopic colorectal surgery: Experience from a non-structured training setting. World J Gastrointest Endosc. 2022 Jun 16;14(6):387-401. doi: 10.4253/wjge.v14.i6.387. PMID 35978712
- [Background] Fox J, Gross CP, Longo W, Reddy V. Laparoscopic colectomy for the treatment of cancer has been widely adopted in the United States. Dis Colon Rectum. 2012 May;55(5):501-8. doi: 10.1097/DCR.0b013e318249ce5a. PMID 22513427